CLINICAL TRIAL: NCT02956083
Title: The Effect of Tear Supplements on Contact Lens Comfort
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of the Incarnate Word (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 14-04-013
Record Dates: First submitted 2016-11-01; First posted 2016-11-04 (Estimated); Last update posted 2016-11-04 (Estimated); Status verified 2016-11

CONDITIONS: Dry Eye Syndromes; Meibomian Gland Dysfunction
MeSH Terms: conditions — Dry Eye Syndromes; Meibomian Gland Dysfunction | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Lipid based artificial tears (Active Comparator): Patients use lipid based artificial tears
  Interventions: Other: Systane Balance eye drops
- Non-lipid based artificial tears (Active Comparator): patients use non-lipid based artificial tears
  Interventions: Other: Systane Contacts eye drops
- Saline (Placebo Comparator): patients use saline
  Interventions: Other: saline

INTERVENTIONS:
Other: Systane Balance eye drops — Propylene Glycol 0.6% Over the counter lipid based artificial tears.
  Arms: Lipid based artificial tears
Other: Systane Contacts eye drops — Hydroxypropyl methycellulose over the counter non-lipid based artificial tears
  Arms: Non-lipid based artificial tears
Other: saline — Saline - no brand name
  Arms: Saline

SUMMARY:
The primary goal of this investigation is to determine if lipid based artificial tear supplementation has an impact on contact lens discomfort (CLD).

DETAILED DESCRIPTION:
Contact lens discomfort (CLD) is the most common cause of discontinuing contact lens wear. Despite years of research and innovations in technology, CLD remains highly prevalent, and thus it is a major concern for patients and practitioners. Studies suggest that meibomian gland dysfunction (MGD) is a cause of CLD. Several lipid-based artificial tears have recently been designed to address dry eye associated with MGD. In this study, the investigators examine if the benefits of lipid based artificial tears extend to improving contact lens comfort. Studies have demonstrated some usefulness of non-lipid based tear supplements in the management of contact lens discomfort. However, the relief was moderate and short-term. To date, no study has examined the impact of lipid based artificial tears on contact lens discomfort. In this study, the investigators will address this gap in knowledge.

ELIGIBILITY:
Inclusion Criteria:

* Patients complaining of contact lens associated discomfort

Exclusion Criteria:

* Patients who do not have contact lens discomfort; patients who have active inflammation or infection of the anterior segment of the eyes.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-07; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Contact Lens Discomfort Questionnaire | 1 months
  CLDEQ Questionnaire will be used to quantify contact lens discomfort

SECONDARY OUTCOMES:
Fluorescein tear break-up time | 1 month
  Fluorescein will be instilled in the conjunctival sac to assess tear break-up time

CONTACTS AND LOCATIONS:
Overall Officials: Srihari Narayanan, OD, PhD, Principal Investigator — University of the Incarnate Word

IPD SHARING:
Plan to Share IPD: No